CLINICAL TRIAL: NCT03439969
Title: The Whole is Greater Than the Sum of Its Parts. "A 8-month Randomised Controlled Trial on the Use of Intra-oral Camera and Text Messages on Gingivitis Control"
Brief Title: A 8-month Study on the Use of Intra-oral Camera and Text Messages on Gingivitis Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lisbon (Other)
Responsible Party: Principal Investigator, Mario Rui Araújo, Master in Health Psychology, University of Lisbon
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Ethic Committee Doc. No. 6/14
Record Dates: First submitted 2018-02-13; First posted 2018-02-20 (Actual); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Behavior and Behavior Mechanisms; Gingivitis
Keywords: Gingivitis; SMS; Text messages; Behavior change; HAPA; Dental Hygiene
MeSH Terms: conditions — Behavior; Gingivitis

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The researcher was blind to the patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (No Intervention): Dental appointment, one hour and included activities that are normally part of a SPT (Suportive Periodontal Treatment) consultation, as well as specific behavior change techniques, such as the use of reinforcement, goal-setting and feedback considered crucial to the accomplishment of long term behavior change. Moreover, special attention was given to patient communication and words such as 'cleaning' and 'hygiene' were replaced by therapeutic synonyms (e.g. inflamed areas and controlling the inflammation) in order to focus patients´ attention on the varied facets of oral health care and increase their perception of the treatment needs. In this group, the device SOPROCARE® by Acteon and Text Messages were not used.
- Intra Oral Camera (Experimental): Dental appointment, one hour and included activities that are normally part of a SPT consultation, as well as specific behavior change techniques, such as the use of reinforcement, goal-setting and feedback. Special attention was given to patient communication and words such as 'cleaning' and 'hygiene' were replaced by therapeutic synonyms (e.g. inflamed areas and controlling the inflammation). In this group, the device SOPROCARE® by Acteon was used in the examination and diagnosis and also for the establishment of therapeutic goals, strategies and skills.
  Interventions: Device: Intra Oral Camera
- Mobile Text Messages (Experimental): Dental appointment, one hour and included activities that are normally part of a SPT consultation, as well as specific behavior change techniques, such as the use of reinforcement, goal-setting and feedback.. Participants in the SMS group further received a total of 16 messages (SMS). One per week.
  Interventions: Device: Mobile Text Messages
- Intra Oral Camera and Text Messages (Experimental): Dental appointment, one hour and included activities that are normally part of a SPT consultation, as well as specific behavior change techniques, such as the use of reinforcement, goal-setting and feedback. Special attention was given to patient communication and words such as 'cleaning' and 'hygiene' were replaced by therapeutic synonyms (e.g. inflamed areas and controlling the inflammation). In this group, the device SOPROCARE® by Acteon was used in the examination and diagnosis and also for the establishment of therapeutic goals, strategies and skills.Participants also received SMS a total of 16 messages (SMS). One per week.
  Interventions: Device: Mobile Text Messages; Device: Intra Oral Camera

INTERVENTIONS:
Device: Mobile Text Messages — Dental inter-proximal control with floss holder and receiving 16 SMS during 4 months.
  Arms: Intra Oral Camera and Text Messages; Mobile Text Messages
Device: Intra Oral Camera — SPT - Appointment with Intra-Oral Camera
  * Examination and diagnosis (15 min) using Intra-oral camera.
  * Motivation, discussion about desired outcomes and treatment needs (using Intra-oral camera) followed by instrumentation (scaling, polishing) (30 min).
  Arms: Intra Oral Camera; Intra Oral Camera and Text Messages

SUMMARY:
To investigate the effects of using an intra-oral camera (IOC) during supportive periodontal therapy, and oral hygiene mobile text messages (SMS) between appointments on clinical, behavioral and psychological parameters of patients with gingivitis.

DETAILED DESCRIPTION:
Dental hygiene behaviours are of paramount importance for controlling gingival health. There is evidence on the use of IOC and of text messages in boosting motivation, sustainability and clinical efficacy of dental hygiene behaviors. Orchestrating these two technologies is expected to create a coaction effect which could improve behavior change interventions, but the effectiveness of such strategy needs to be inspected.

ELIGIBILITY:
Inclusion Criteria:

Gingivitis BOMP > 0.5 20 teeth (minimum 5 per quadrant) > 18 years old

Exclusion Criteria:

periodontitis (pockets >3), smoking, orthodontics, pregnancy removable partial dentures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 233 (Actual)
Dates: Start 2014-06-01 (Actual); Primary Completion 2015-02-28 (Actual); Study Completion 2016-11-30 (Actual)

PRIMARY OUTCOMES:
Change from BOMP (Bleeding on Marginal Probing) at 4 & 8 months | Baseline, 4 months & 8 months
  Gingival bleeding Index

SECONDARY OUTCOMES:
HAPA (Health Action Process Approach) behavioral variables questionnaire. | Baseline, 4 & 8 months.
  Measures adapted to oral health from previous studies with the HAPA model (Godinho et al. 2015) were used. All the HAPA variables were evaluated using a 7 point Likert-type scale, ranging from totally disagree (1) to totally agree (7), unless otherwise stated.
SMS (Short Messages Service) text messages opinion questionnaire | At 4 months.
  Opinion about receiving SMS and how can it influence the appointment.
Intra Oral Camera opinion questionnaire | At 4 and 8 months.
  Opinion about receiving Intra Oral camera and how can it influence the appointment.
Self-report Dental Hygiene Behaviors questionnaire. | Baseline, 4 and 8 months.
  Level of toothbrushing and dental floss frequency.

REFERENCES:
- [Background] Godinho CA, Alvarez MJ, Lima ML, Schwarzer R. Health messages to promote fruit and vegetable consumption at different stages: A match-mismatch design. Psychol Health. 2015;30(12):1410-32. doi: 10.1080/08870446.2015.1054827. Epub 2015 Jul 24. PMID 26010304